CLINICAL TRIAL: NCT03941171
Title: The Effect of PAO Followed by Progressive Resistance Training Versus Progressive Resistance Training in Patients With Hip Dysplasia. A Randomized Controlled Trial
Brief Title: Is Periacetabular Osteotomy Superior to Progressive Resistance Training?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); VIA University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PreserveHIP
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Hip Dysplasia
Keywords: Periacetabular Osteotomy; Progressive resistance training; PAO
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): PAO+usual+PRT
  Interventions: Procedure: PAO; Other: Usual care after PAO; Other: PRT
- Group 2 (Active Comparator): PRT
  Interventions: Other: PRT

INTERVENTIONS:
Procedure: PAO — PAO will be performed as the trans-sartorial approach or the anterior pelvic approach.
  Arms: Group 1
Other: Usual care after PAO — Patients commence post-operative rehabilitation as usual and follow the rehabilitation program guided by a physiotherapist specialized in hip problems until 4 months after the operation.
  Arms: Group 1
Other: PRT — 4 months of partly supervised progressive resistance training 2 times per week. After these 4 months (16 weeks), patients receive a free membership to a fitness center near their home address and are encouraged to train on their own 2 times per week until 12 months follow-up with one supervised session per month. The PRT program involves 10-min of warm up followed by 50-min of bilateral resistance exercises including sets of squats, hip extension, hip flexion, and hip abduction.

SUMMARY:
The primary aim of this study is to examine if Periacetabular Osteotomy (PAO) followed by 4 months of usual care followed by 8 months of progressive resistance training (PRT) is superior to 12 months of a PRT intervention in patients with hip dysplasia eligible for PAO in terms of self-reported pain on the HAGOS questionnaire. Secondary aims are to investigate changes in patient-reported symptoms, physical function in daily living, physical function in sport and recreation, hip and/or groin-related quality of life, generic health status, functional performance, muscle strength, physical activity and adverse events between PAO followed by usual care+PRT compared to PRT only. We hypothesise that in patients with hip dysplasia, PAO followed by usual care+PRT, results in significantly less pain at 12 months follow-up, compared to PRT only.

DETAILED DESCRIPTION:
Group 1 (PAO+usual+PRT):

PAO will be performed as the trans-sartorial approach or the anterior pelvic approach. Patients commence post-operative rehabilitation as usual and follow the rehabilitation program guided by a physiotherapist specialized in hip problems until 4 months after the operation. 4 months postoperative the patients complete usual care and continue with the same PRT intervention program as the PRT group, with 4 months of supervised sessions (see description below).

Group 2 (PRT):

The PRT group receives 4 months of supervised PRT 2 times per week. A physiotherapist or students will supervise all training sessions the first 4 weeks. The following 4 weeks, 6 out of 8 training sessions are supervised and from week 9-16, half of the training sessions (8 out of 16) are supervised. After these 4 months (16 weeks), patients receive a free membership to a fitness center near their home address and are encouraged to train on their own 2 times per week until 12 months follow-up with one supervised session per month. The PRT program involves 10-min of warm up followed by 50-min of bilateral resistance exercises including sets of loaded squats, hip extension, hip flexion, and hip abduction. The absolute training load will be individually adjusted on a set-by-set basis, using the plus two principle (if the patient is able to perform two or more repetitions than required, the load is increased). Hip related pain levels up to 5 on the VAS is considered acceptable during exercise.

The study is a multicentre randomised controlled and assessor blinded trial. Primary endpoint will be 12 months after initiation of surgical/non-surgical treatment. Secondary endpoints will be measured at 4 months after the start of the treatment (surgical/non-surgical). In addition, 5-year and 10-year follow-up with questionnaires is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-45 years and diagnosed with hip dysplasia referred from primary care to the Department of Orthopaedic Surgery at one of the two participating hospitals.
2. Considered eligible for PAO by a surgeon.
3. Radiographic verified hip dysplasia (CE-angle <25 degrees and AI-angle >10 degrees) and clinical symptoms.
4. Range of motion: internal rotation >15 degrees, external rotation >15 degrees, hip flexion >110 degrees.
5. Able to commute to training sessions.

Exclusion Criteria:

1. OA degree ≥1 on classification of Tönnis'.
2. CE-angle <10 degrees.
3. Previous pelvic surgery for hip dysplasia (affected side).
4. Calvé Legg Perthes or epifysiolysis.
5. Simultaneous bilateral PAO.
6. Previous surgery for herniated disc, spondylodesis, arthroplasty of hip, knee or ankle.
7. Previous surgery of the hip (tenotomy of iliopsoas tendon, z-plastic of the iliotibial tract or hip arthroscopy) in index leg.
8. Neurological or rheumatoid diseases that affect the hip function.
9. Inadequacy in written and spoken Danish or Norwegian.
10. Body Mass Index (BMI) >25 in Aarhus and BMI >30 in Oslo and Odense

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in pain related to hip function, between baseline and 12 months follow-up | Measured at baseline, 4 month follow-up and 12 month follow-up
  The pain subscale of the patient reported questionnaire Copenhagen Hip and Groin Outcome Score (HAGOS), were the total score ranges from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Change in self-reported hip function | Measured at baseline, 4 month follow-up and 12 month follow-up
  The subscales; Symptoms, Physical function in daily living, Physical function in Sport and Recreation, Participation in Physical Activities and hip and/or groin-related Quality of Life of the patient reported questionnaire Copenhagen Hip and Groin Outcome Score (HAGOS), where the total score ranges from 0 (worst) to 100 (best).
Change in hip function | Measured at baseline, 4 month follow-up and 12 month follow-up
  Single leg hop for distance is a test that measure functional performance requiring both strength, power and balance. The distance from start to landing is measured in cm. and height adjusted by dividing the distance of the hop with the height of the patient.
Change in balance function | Measured at baseline, 4 month follow-up and 12 month follow-up
  The Y balance test require strength, flexibility, neuromuscular control, stability, range of movement, balance and proprioception. These elements are tested and the maximal reach distance is recorded for each direction (anterior, posteromedial and posteroladeral). The composite reach is calculated and normalized to limb length for analysis of the overall performance on the test.
Number of patients with adverse events and serious adverse events after PAO | Reported within 12 months after surgery
  Adverse events:
  * Haematoma
  * Delayed wound closure
  * Dysaethesia of lateral femoral cutaneous nerve
  * Malpositioning; retroversion or insufficient reorientation. Insufficient reorientation (coverage) - optimal is CE angle 30-40 degrees. AI angle 0-10 degrees.
  * Heterotopic ossifications (Brooker I and II)
  * Urinary tract infections
  * Infection not requiring surgical revision
  Serious adverse events:
  * Avascular necrosis of the femoral head or acetabulum
  * Nerve palsy
  * Major bleeding (administration of more than 5 blood units intra- and postoperatively)
  * Peroneal and femoral neurapraxia
  * Deep vein thrombosis
  * Pulmonary embolism
  * Stress fracture of ischial bone and posterior column
  * Intraarticular osteotomy
  * Heterotopic ossifications (Brooker III and IV)
  * Infection requiring surgical revision
  * Loss of fixation/loss of reorientation
  * Delayed or non-union of pubic, ischial or iliac bone
Change in usage of painkillers | Measured at baseline, 4 month follow-up and 12 month follow-up
  Usage of painkillers (yes/no), including type of painkillers (Paracetamol, NSAID, Morfin/opiods and/other type of medicine)
Change in self-reported pain | Measured at baseline, 4 month follow-up and 12 month follow-up
  Pain reported by the Visual Analogue Scale (VAS). A scale where pain is marked from 0-100, and 0 is no pain and 100 is worst imaginable pain.
Change in hip awareness | Measured at baseline, 4 month follow-up and 12 month follow-up
  Hip awareness is measured with the Forgotten Joint Score questionnaire (FJS), where each patient completes the 12 questions regarding awareness of their affected hip. Each question is answered with one of the following options; never, almost never, seldom, sometimes and mostly, corresponding to a score of 1-5. The sum of the scores will be converted into a score between 0-100. A high score will indicate lack of awareness and a low score will indicate great awareness of the affected hip.
Change in muscle strength | Measured at baseline, 4 month follow-up and 12 month follow-up
  Muscle strength in hip-abduction, hip-flexion and hip-extension is measured isometrically, with a dynamometer.

OTHER OUTCOMES:
Change in physical activity | Measured at baseline and 12 month follow-up
  Tri-axial accelerometer
Change in patient-reported health | Measured at baseline, 4 month follow-up and 12 month follow-up
  Change in patient-reported health will be measured with the EuroQol Group 5-dimension patient-reported questionnaire (EQ-5D-5L), where each dimension has five response levels; ranging from no problems to extreme problems (level 1 to level 5). The scores will be combined, using one level from each dimension, ranging from 11111 (best health) to 55555 (worst health). The instrument also includes a visual analogue scale (VAS) where self-perceived health is scored on a 0 to 100 mm scale representing "the worst health you can imagine" and "the best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Lisa U Tønning, MSc, Principal Investigator — Department of Orthopedic Surgery, Aarhus University Hospital, Denmark; Inger Mechlenburg, DMSc, PhD, Study Director — Department of Clinical Medicine, Aarhus University, Denmark; Ulrik Dalgas, MSc, PhD, Study Director — Department of Public Health - Sport, Aarhus University, Denmark; Stig S Jakobsen, PhD, Study Director — Department of Orthopedic Surgery, Aarhus University Hospital, Denmark; Kjeld Søballe, DMSc, Study Director — Department of Orthopedic Surgery, Aarhus University Hospital, Denmark; Julie S Jacobsen, MSc, Study Director — Department of Physiotherapy & Research Centre in Health and Welfare Technology, VIA University College, Denmark; Jan E Madsen, MD, PhD, Study Director — Department of Orthopedic Surgery, Oslo University Hospital, Norway; Lars Nordsletten, PhD, Study Director — Division of Orthopaedic Surgery, Oslo University Hospital, Oslo; Faculty of Medicine, University of Oslo, Norway; Tone Bere, PT, PhD, Study Chair — Department of Orthopedics, Oslo University Hospital Ullevaal, Norway; May A Risberg, PhD, Study Director — Department of Orthopedics, Oslo University Hospital Ullevaal, Norway
Locations (3):
- Denmark (2):
  - Lisa Urup Tønning, Aarhus N, Central Jutland
  - Odense University Hospital, Odense, Fyn
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Aarhus University Hospital is responsible for handling all personal data provided by both sites in accordance to the Clinical Trial Agreement and the EU General Data Protection Regulation (GDPR).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: End of study and 5 years ahead
Access Criteria: Oslo University Hospital agree that information directly related to the protocol and trial, including data, material, Intellectual Property and results generated from the trial shall be the property of Aarhus University Hospital, and shall be treated in strict confidence, and shall not be disclosed to any third party, or use for its benefit or the benefit of any third party, without the prior written consent of Aarhus University Hospital, except for data that is (i) publicly known or available from other sources who are not under a confidentially obligation to the other party; (li) has been made available by the other party without confidentiality obligation; or (iii) is independently developed or otherwise already known by or available to the other party without a confidentiality obligation; or (iv) is already required disclosed by law.

REFERENCES:
- [Derived] Reimer LCU, Jakobsen SS, Mortensen L, Dalgas U, Jacobsen JS, Soballe K, Bere T, Madsen JE, Nordsletten L, Risberg MA, Mechlenburg I. Efficacy of periacetabular osteotomy followed by progressive resistance training compared to progressive resistance training as non-surgical treatment in patients with hip dysplasia (PreserveHip) - a protocol for a randomised controlled trial. BMJ Open. 2019 Dec 23;9(12):e032782. doi: 10.1136/bmjopen-2019-032782. PMID 31874882

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT03941171/Prot_SAP_000.pdf